CLINICAL TRIAL: NCT04328506
Title: Randomized,Open Label,Two-cycle,Crossover,Single Dose Bioequivalency Study of Two Preparations of CM082 Tablet in Healthy Chinese Volunteers Under Fasted State and After Meal
Brief Title: Bioequivalency Study of CM082 Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-108
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2020-03

CONDITIONS: Advanced Malignant Solid Tumors
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T-R cohort under fasted state (Experimental): Subjects will be administered with one single dose of CM082 tablet (test product) under fasted state, after a wash period of 5 days, the subjects will be administered with one single dose of CM082 tablet (reference product) under fasted state.
  Interventions: Drug: CM082 tablet (test product); Drug: CM082 tablet (reference product)
- R-T cohort under fasted state (Experimental): Subjects will be administered with one single dose of CM082 tablet (reference product) under fasted state, after a wash period of 5 days,the subjects will be administered with one single dose of CM082 tablet (test product) under fasted state.
  Interventions: Drug: CM082 tablet (test product); Drug: CM082 tablet (reference product)
- T-R cohort after meal (Experimental): Subjects will be administered with one single dose of CM082 tablet (test product) after meal, after a wash period of 5 days,the subjects will be administered with one single dose of CM082 tablet (reference product) after meal.
  Interventions: Drug: CM082 tablet (test product); Drug: CM082 tablet (reference product)
- R-T cohort after meal (Experimental): Subjects will be administered with one single dose of CM082 tablet (reference product) after meal, after a wash period of 14 days,the subjects will be administered with one single dose of CM082 tablet (test product) after meal
  Interventions: Drug: CM082 tablet (test product); Drug: CM082 tablet (reference product)

INTERVENTIONS:
Drug: CM082 tablet (test product) — Test product(T)：100mg CM082 tablet manufactured by Betta Pharmaceuticals
Drug: CM082 tablet (reference product) — Reference product(R)：100mg CM082 tablet manufactured by Catalent Pharma Solutions

SUMMARY:
The main objective of this study is to evaluate the bioequivalency of two preparations of CM082 tablet in Chinese healthy volunteers.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the bioequivalency of two preparations of CM082 tablet in Chinese healthy volunteers under fasted state or after meal. In addition, the safety of single dose administration of CM082 tablet in Chinese healthy volunteers will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male body weight≥50.0kg or female body weight≥45.0kg; BMI between 19.0-26.0 kg/m2(inclusive)
* Generally in good health, with no history of chronic disease or sever disease
* No (clinical significant) abnormal findings in clinical laboratory tests and physical examinations
* No plan for pregnancy in coming 6 months, and must practice effective contraception; No plan for sperm or egg donation
* Written informed consent

Exclusion Criteria:

* History of food or drug allergies
* Clinical significant disease or disorders
* Received surgery in 3 months before screening, or have plan for surgery during the study
* Participated in other clinical trials within 3 months before screening
* Intolerant of venipuncture, history of fainting needle and blood
* Lactose intolerant
* Drug abusing in 3 months
* Donated ≥200 mL of blood within 3 months before screening
* Pregnant or under lactation period (female subjects)
* Received any prescription drug, over-the-counter drug, prescription drug and Chinese herbal drug in 2 weeks, with the exception of vitamins and acetaminophen
* Received any vaccine in 4 weeks
* Excessively smoking, alcohol or coffin-containing beverage drinking in 3 months
* Other circumstances that is deemed not appropriate for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration(Cmax) of CM082 (test product or reference product) under fasted state or after meal | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,7,8,10,12,16,24,36,48,72 hour]
  The Cmax ofCM082 (test product or reference product) in under fasted state or after meal blood samples of each subject over a 72 hour period post dose
Area under the plasma concentration versus time curve(AUC) of CM082 (test product or reference product) under fasted state or after meal | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,7,8,10,12,16,24,36,48,72 hour]
  The AUC of CM082 (test product or reference product) in under fasted state or after meal blood samples of each subject over a 72 hour period post dose
Time of maximum concentration (Tmax) of CM082 (test product or reference product) under fasted state or after meal | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,7,8,10,12,16,24,36,48,72 hour]
  The Tmax of CM082 (test product or reference product) in under fasted state or after meal blood samples of each subject over a 72 hour period post dose

SECONDARY OUTCOMES:
Percentage of adverse events | From the first occurrence of adverse events after administration to the cessation of adverse events, assessed up to 2 months
  Percentage of adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: zourong ruan, Study Chair — the Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- The 1st Phase Clinical Research Center of the Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China